CLINICAL TRIAL: NCT06489470
Title: Strokectomy in Malignant Cerebral Media Infarction: A Pilot Study
Brief Title: Strokectomy in Malignant Cerebral Media Infarction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rostock (Other)
Responsible Party: Principal Investigator, Sae-Yeon Won, Associate Professor, University of Rostock
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMR1
Record Dates: First submitted 2024-06-26; First posted 2024-07-08 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Stroke, Ischemic
Keywords: necrosectomy; alternative surgical treatment; strokectomy
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Necrosectomy/Strokectomy (Experimental)
  Interventions: Procedure: Strokectomy/Necrosectomy

INTERVENTIONS:
Procedure: Strokectomy/Necrosectomy — After obtaining CT-/MRT-perfusion, the infarcted area (e.g. infarct core) of malignant MCA-infarction is localized. By using the neuronavigation, surgical resection of necrotic tissue is performed in a non-eloquent area until the space occupying effect is released. At the end of the surgery, the bone flap is reinserted and fixated.

SUMMARY:
Decompressive hemicraniectomy (DC) is the standard procedure and life saving measure in case of malignant middle cerebral artery (MCA) infarction. However, there have been several studies reporting the neuroinflammatory cascade based on the necrotic tissue as one of the leading cause for the secondary brain damage, wherefore, strokectomy with resection of necrotic tissue has been proposed in some case series as an alternative surgical option. Thus, the aim of this study is to perform a pilot study by including patients with malignant MCA infarction and to check the feasibility of this specific surgical treatment.

DETAILED DESCRIPTION:
Ischemic stroke is one of the leading causes of disability and death worldwide. While cerebral middle cerebral artery (MCA) infarction constitutes approximately 10% of all ischemic, it is a life-threatening medical emergency causing a mass effect with substantial rise in intracranial pressure and reduction of cerebral blood flow. The letality of malignant MCA-infarction under conservative treatment lies around 70%, wherefore a surgical treatment is important in these patients. In the past years, there have been several randomized controlled trials (DESTINY, DECIMAL, HAMLET) focussing on the decompressive hemicraniectomy (DC) in malignant MCA infarction. Those studies have shown the superiority of DC compared to medical management in higher rate of survival and favorable outcome measured by modified Rankin Scale (mRS). Consequently, the DC is recommended as a life-saving treatment in the American Stoke Association for patients under 60 years of age. Further, the DESTINY II trial could show the beneficial effect of DC in patients over 60 years of age as well, wherefore the age alone is not a cut-off line anymore to indicate a surgical treatment.

Despite this life saving measure, there are several sequelae of DC to consider. Patients who have survived usually undergo a second surgery to close the skull defect by cranioplasty. As previous study reported, the surgical procedure of cranioplasty inherits a high complication rate up to 34% including infection, wound impairment, intracranial hemorrhage and aseptic necrosis. Further, DC can cause a syndrome of the trephined or hydrocephalus which is associated with additional risk for patient and increased cost for the community.

Recently, investigator´s research group performed a multicentric study across academic hospitals in Germany including over 500 patients with cerebellar infarction. As a subgroup analysis, investigators compared the functional outcome in these cohorts considering different surgical treatment strategies: craniotomy+necrosectomy versus DC. According to this study, craniotomy + necrosectomy was superior in higher rate of favorable outcome at discharge and at 3 months follow-up compared to DC. This result is supported by a recent systematic review and meta-analysis by Ayling et al. as well. In line with this, resection of infarcted frontal/temporal lobe has been proposed as surgical alternative to DC in malignant MCA-infarction (defined as "strokectomy", "necrosectomy"). In a recent systematic review and meta analysis, there was a clear trend towards higher favorable outcome in necrosectomy group compared to DC group (mRS 0-3: 58.5% vs 39.4%) with malignant MCA-infarction, however, further clinical studies are needed for more evidence concerning the specific surgical method to integrate in the clinical routine.

Pathophysiologically, it has been shown that the neuroinflammatory cascade ensue during ischemic stroke. Experimental and clinical studies support the existence of inflammatory area surround the initial lesion in the subacute phase of ischemic stroke, which was defined as "inflammatory penumbra". Cellar death occurs in this region with triggering cytotoxic T-cells resulting in increased cell death and cytotoxic edema. This phenomenon might have contributed to the superior functional results observed in the necrosectomy group in ischemic stroke, but this hypothesis has to be proved in the future studies.

Thus, the general aims are to evaluate the functional outcome of malignant MCA-infarction treated either by necrosectomy or DC in an international, multicentric large cohort of patients. Prior to this study, the aim of current study is to perform a pilot study performing necrosectomy in malignant MCA-infarction to proof the feasibility of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Ischemic middle cerebral artery (MCA) infarction at least two thirds of the MCA territory
* Clinical symptoms of acute unilateral MCA infarction less than 48 hours prior to the initiation of treatment

Exclusion Criteria:

* Preexisting modified Rankin Scale >2
* Absence of pupillary reflexes or GCS <6
* Intracerebral hemorrhage or other associated brain lesions
* Contraindications for surgery
* Estimated life expectancy of less than 3 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-06-15 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Rate of resurgery after necrosectomy of malignant MCA-infarction | up to 2 weeks
  After the surgical treatment, the patients will be treated in the neurointensive care unit. During the clinical course, the necessity to perform a secondary surgery (e.g. hemicraniectomy) will be observed. For the safety of the patients, intracranial pressure monitoring will be continously performed as well.

SECONDARY OUTCOMES:
Surgical complications | up to 3 months
  The rate of wound infection, other infections, postoperative hemorrhage and postoperative seizure will be documented during the clinical course and follow-up.
Functional outcome via modified Rankin Scale (mRS; range 0-6; 0-3: favorable outcome, 4-6: unfavorable outcome) at 3 months | up to 3 months
  After 3 months, the functional outcome will be evaluated by modified Rankin Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Sae-Yeon Won, MD, Principal Investigator — Neurosurgery, University Medical Center Rostock; Florian Gessler, MD PhD, Study Director — Neurosurgery, University Medical Center Rostock; Matthias Wittstock, MD, Study Chair — Neurology, University Medical Center Rostock
Locations (1):
- University Medical Center Rostock, Rostock, Mecklenburg-Vorpommern, Germany

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Up to 12 months